CLINICAL TRIAL: NCT02026570
Title: Enhancement of Residual Limb Proprioception and Rehabilitation Training Methods With a Vibrotactile Device.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Southern California Institute for Research and Education (Other)
Collaborators: California State University, Long Beach (Other); California State University, Dominguez Hills (Other)
Responsible Party: Principal Investigator, Dana Craig, Health System Specialist, Southern California Institute for Research and Education
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 01234
Record Dates: First submitted 2013-12-19; First posted 2014-01-03 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Transtibial Amputation
Keywords: Prosthesis; Falls; Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Persons with unilateral transtibial amputation receiving standard physical therapy.
- Motor Control Internal Focus (Experimental): Persons with unilateral transtibial amputation receiving standard physical therapy and additional training with motor control internal focus of attention instructions.
  Interventions: Behavioral: Internal Focus of Attention
- Motor Control External Focus (Experimental): Persons with unilateral transtibial amputation receiving standard physical therapy and additional training with external focus of attention instructions.
  Interventions: Behavioral: External Focus of Attention

INTERVENTIONS:
Behavioral: Internal Focus of Attention — Providing instructions for the user to manipulate their residual limb in space during standing and walking tasks.
  Arms: Motor Control Internal Focus
Behavioral: External Focus of Attention — Providing instructions for the user to manipulate their prosthetic foot in space during standing and walking tasks.
  Arms: Motor Control External Focus

SUMMARY:
Objectives: The purpose of this study is to investigate attentional (internal vs. external) focus effects on persons with amputation to perform a defined compensatory movement to reduce the likelihood of a fall. An internal focus of attention directs a person's conscious attention to their body's movements, whereas an external focus of attention directs a person's conscious attention to the effects of their movements or specific features in the environment. Numerous experiments have investigated the effects of an internal and external focus of attention on motor performance and the findings are in favor of an external focus of attention. In our work, we propose a motor learning research experiment to evaluate attentional focus strategies on the rehabilitation outcomes of learning and adaptation to the new proprioceptive information for persons with a recent transtibial amputation.

Research Design and Methodology: For this pilot study, six participants with recent unilateral transtibial amputation will be recruited. Four participants will receive internal and external focus of attention training methods while the other two (control group) will receive standard prosthetic training instructions. The experiment will be conducted in three phases: Phase 1 -- Baseline Performance Test, Phase 2 -- Training sessions, and Phase 3 - Learning Test. The training will utilize a vibrotactile device designed to generate tactile sensations at the skin-socket interface simulating contact of the prosthesis with the environment. The sensation simulates a perturbation that signals a potential fall event. During the experiment the augmented sensory information will be introduced randomly while participants walk at a preferred pace on a level surface. Movement kinematics and kinetics of the body will be recorded for analyses using a motion capture system with force plates.

Finding: It is hypothesized that the external focus of attention condition will outperform the internal focus of attention condition when responding to perturbations. The external focus of attention condition will yield faster response time and show improved compensatory responses compared to the internal focus of attention group by producing a greater lateral displacement of the artificial limb relative to the line of progression. In addition, the external condition will demonstrate a greater step length and step height than the internal focus of attention condition when provided with a perturbation.

Clinical Significance: Current practices within the field of Physical Therapy reveal that there is little therapeutic intervention for fall prevention. Instructions are traditionally provided on how to reduce the risk of falling through preparation of a room or obstacle avoidance or on the proper way to fall to decrease injury. However, there are no protocols for providing a prosthetic user with compensatory strategies to avoid a fall after a perturbation occurs. The research findings can result in improved training protocols, which can improve rehabilitative outcome.

Impact/Significance: The growing number of prosthetic users presents a need for improved patient care and effective prosthetic training and rehabilitation methods. Complimentary to the mission of the VA, the results of this research could enhance the quality of patient care and further assist these patients toward becoming prosthetically rehabilitated.

ELIGIBILITY:
Inclusion Criteria:

* Undergone amputation within the past year.
* Currently undergoing prosthetic training in Physical Therapy utilizing a prosthesis.
* Be within two weeks of completing prosthetic training in Physical Therapy.
* Ability to tolerate walking for a minimum of 100 yards over the course of a four hour time period with or without resting.
* No current skin breakdown on the residual limb.

Exclusion Criteria:

* Not cleared by Physical Therapy to use the prosthesis without contact precautions.
* Any medical or psychosocial condition that, in the opinion of the investigator, could jeopardize the subject's participation, and compliance with the study criteria

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2013-06 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Reaction Time | Five visits over a three week period.
  Time for subject to laterally displace Center of Mass two standard deviations from normative trajectory following stimulus.

SECONDARY OUTCOMES:
Movement Time | Five visits over a three week period.
  Time from reaction time to completion of task, which is a side step following stimulus.

CONTACTS AND LOCATIONS:
Overall Officials: Dana D. Craig, M.A., Principal Investigator — V.A. Long Beach Healthcare System
Locations (1):
- V.A. Long Beach Healthcare System, Long Beach, California, United States

REFERENCES:
- [Background] Clippinger FW, Seaber AV, McElhaney JH, Harrelson JM, Maxwell GM. Afferent sensory feedback for lower extremity prosthesis. Clin Orthop Relat Res. 1982 Sep;(169):202-6. PMID 7105581
- [Background] D. J. DiLorenzo, D. J. Edell, M. J. Koris, and R. R. Riso, "Chronic intraneural electrical stimulation for prosthetic sensory feedback," 1st IEEE EMBS Conference on Neural Engineering, pp:116-119, 2003.
- [Background] Doubler JA, Childress DS. An analysis of extended physiological proprioception as a prosthesis-control technique. J Rehabil Res Dev. 1984 May;21(1):5-18. PMID 6527290
- [Background] Fan RE, Culjat MO, King CH, Franco ML, Boryk R, Bisley JW, Dutson E, Grundfest WS. A haptic feedback system for lower-limb prostheses. IEEE Trans Neural Syst Rehabil Eng. 2008 Jun;16(3):270-7. doi: 10.1109/TNSRE.2008.920075. PMID 18586606
- [Background] Kaczmarek KA, Webster JG, Bach-y-Rita P, Tompkins WJ. Electrotactile and vibrotactile displays for sensory substitution systems. IEEE Trans Biomed Eng. 1991 Jan;38(1):1-16. doi: 10.1109/10.68204. PMID 2026426
- [Background] Kadkade PP, Benda BJ, Schmidt PB, Wall C 3rd. Vibrotactile display coding for a balance prosthesis. IEEE Trans Neural Syst Rehabil Eng. 2003 Dec;11(4):392-9. doi: 10.1109/TNSRE.2003.819937. PMID 14960115
- [Background] G.E. Loeb and F.J. Richmond. BION Implants for Therapeutic and Functional Electrical Stimulation. Neural Prostheses for Restoration of Sensor and Motor Function. CRC Press, Boca Raton, FL, 2000. R.A. Magill. "Motor Learning and Control: Concepts and Applications," (9th ed.). New York, NY: McGraw Hill, 2011
- [Background] Miller WC, Speechley M, Deathe B. The prevalence and risk factors of falling and fear of falling among lower extremity amputees. Arch Phys Med Rehabil. 2001 Aug;82(8):1031-7. doi: 10.1053/apmr.2001.24295. PMID 11494181
- [Background] J.A. Sabolich and G.M. Ortega. "Sense of feel for lower-limb amputees: A phase-one study," Journal of Prosthetics and Orthotics, 6(2):36-41, 1994
- [Background] J.A. Sabolich, G.M. Ortega, and G.B. Schwabe. "System and method for providing a sense of feel in a prosthetic or sensory impaired limb," United States Patent, December 31, 2002
- [Background] D.C. Simpson. "The choice of control system for the multimovement prosthesis: extended physiological proprioception (EPP), " In: The Control of Upper-Extremity Prostheses and Orthoses. Springfiled, Illinois, C.C Thomas. pp:146-150, 1974
- [Background] D.C. Simpson. "The control and supply of a multimovement externally powered upper limb prosthesis," Proc 4th Ini Symp External Control of Human Extremities. Belgrade, Yugoslav Committee for Electronics and Autotlon. pp:247-254, 1973
- [Background] Wulf G, Prinz W. Directing attention to movement effects enhances learning: a review. Psychon Bull Rev. 2001 Dec;8(4):648-60. doi: 10.3758/bf03196201. PMID 11848583
- [Background] Yoshida K, Horch K. Closed-loop control of ankle position using muscle afferent feedback with functional neuromuscular stimulation. IEEE Trans Biomed Eng. 1996 Feb;43(2):167-76. doi: 10.1109/10.481986. PMID 8682528
- [Background] D. Zambarbieri, M. Schmid, and G. Verni. "Sensory feedback for lower limb prosthesis", in Intelligent Systems and Technologies in Rehabilitation Engineering, Ed. H.L. Teodorescu and L. Jain, CRC Press, Boca Raton, 2001